CLINICAL TRIAL: NCT05126875
Title: Re-TREAT: A Phase 2 Study of Stereotactic Re-irradiation of Relapsed Brain Metastases
Brief Title: Re-TREAT: Re-irradiation for Relapsed Brain Metastases
Acronym: RE-TREAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Søren Møller, MD, Consultant, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RE-TREAT
Record Dates: First submitted 2021-08-09; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Cancer; Brain Metastases, Adult
MeSH Terms: conditions — Neoplasms; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Treatment with stereotactic radiosurgery
  Interventions: Radiation: Repeated stereotactic radiosurgery

INTERVENTIONS:
Radiation: Repeated stereotactic radiosurgery — Repeated stereotactic radiosurgery to recurring brain metastases
  Other Names: SRS

SUMMARY:
The Re-TREAT study is a prospective clinical, phase 2, interventional, single-arm, multicenter trial for patients with local relapse of one or more brain metastases. Patients with recurrence of one or more brain metastases that have previously been treated with stereotactic radiosurgey (SRS) are treated with repeated SRS. The aim is to evaluate the efficacy and toxicity of salvage SRS. The primary outcome is local control of the relapsed tumor and the secondary endpoints include toxicity as evaluated by the investigator and quality of life measured as a patient reported outcome. As an exploratory endpoint, the value of advanced MRI (magnetic resonance imaging) and PET (positron emission tomography) imaging as a biomarker for prediction of response to treatment or toxicity will be studied.

DETAILED DESCRIPTION:
Background It is estimated that 10-20 % of patients with cancer develop brain metastases (BM) and the number is increasing due to prolonged patient survival as a result of improvements in surgery and systemic treatment. With few exceptions however, chemotherapy is not effective in treating disease within the central nervous system and therefore BM are often treated as a separate compartment independently from the rest of the disease throughout the body. Treatment modalities include surgical resection, stereotactic radiosurgery (SRS) and whole brain irradiation (WBI) or a combination.

SRS is a technique where a high dose of radiation is delivered through multiple fields, often as rotational intensity modulated radiation therapy (IMRT), where the beam is aimed at the tumor from everchanging angles, in order to minimize the dose to the surrounding tissue. In contrast to other radiation modalities, where a margin is added to the target in order to eradicate tumor cells that are not visible on imaging, SRS employs very small margins because brain metastases tend to be localized with sharp boundaries to surrounding tissue. The relative low dose absorbed by the surrounding tissue allows for delivery of the whole radiation dose to the tumor in one to three treatment sessions ('fractions'), as opposed to conventionally fractionated radiotherapy which is delivered in multiple fractions for the protection of surrounding healthy tissue.

As a whole, SRS results in high rates of local tumor control (65-90%) and low rates of toxicity (10-15%), which is usually mild. The most significant adverse event following SRS is radionecrosis, which is estimated to occur in 5-25% of patients. This is a condition which is poorly defined but is commonly used to describe a situation where the contrast enhancing area in the irradiated volume increases, often accompanied by increasing edema in the surrounding tissue. The condition may or may not cause symptoms. In cases of symptomatic, progressive radionecrosis, oral corticosteroids such as prednisolone may be needed for longer periods of time. Differentiation between relapsed metastasis and radionecrosis is notoriously difficult and represents one of the major diagnostic challenges in all of neuro-oncology. Advanced imaging techniques such as dynamic MRI (e.g. perfusion weighted images) or PET (positron emission tomography) have been used to aid in differentiation in experimental studies, but this currently remains an area of research. The development of the brain lesion over time and use of close follow-up using MRI will most often aid in interpretation of the images by the multidisciplinary team conference consisting of a radiologist, a radiation oncologist and a neurosurgeon.

There is no standard treatment in case of local tumor relapse following SRS. Patients who have not previously received WBI may be offered this, but the possible detrimental effects on neurocognition and quality of life are well documented4 and many clinicians as well as patients prefer to avoid this for as long as possible. Few patients in this category are recommended surgical resection.

Salvage SRS (repeated SRS to the same area at time of relapse) is commonly practiced at some institutions, Rigshospitalet being one of them, but the evidence to support routine use is sparse. The treatment has been evaluated only in retrospective studies. These have found high rates of local control (70-90%), but as adverse events and side effects cannot be evaluated from retrospective studies without risk of critical bias, the safety of this treatment remains to be established.

Aim of the study The Re-TREAT study is a prospective clinical, phase 2, interventional, single-arm, multicenter trial with patients with local relapse of one or more brain metastases. In the trial, they are treated with salvage SRS. The aim is to evaluate the efficacy and toxicity of salvage SRS. The primary outcome is local control of the relapsed tumor and the secondary endpoints include toxicity as evaluated by the investigator and quality of life measured as a patient reported outcome. As an exploratory endpoint, the value of advanced MRI and PET-imaging as a biomarker for prediction of response to treatment or toxicity will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Brain metastases of solid tumor (carcinoma of unknown origin may be included but histological verification in case of BM alone is required)
* Progression of previously treated lesion as decided by the multidisciplinary team conference
* Previous single fraction SRS in area in question and dose plans must be available electronically
* Previous single fraction SRS given > 3 months previously
* ECOG (Eastern Cooperative Oncology Group) performance status ≤2
* Life expectancy >3 months
* Signed written consent.
* Patients may have more than one recurring lesion and may also have new, untreated metastases which may be treated with standard SRS (up to a total of 4 metastases in accordance with Danish national guidelines).

Exclusion Criteria:

* Two previous courses of radiotherapy for the same metastasis (e.g. SRS and WBRT)
* Target lesions located in- or in proximity to eloquent brain areas that require reduction of radiotherapy dose
* Target lesion gross tumor volume (GTV) for radiotherapy greater than 14,1 cm3 (equivalent to a sphere with a diameter of 3 cm)
* Current or planned concomitant medical treatment that is likely to be active against brain metastases (e.g. tyrosine kinase inhibitors for EGFR-positive (epidermal growth factor receptor) non-small cell lung cancer) or that may influence interpretation of images (e.g. bevacizumab, a monoclonal antibody directed towards VEGF (vascular endothelial growth factor)) in the opinion of the investigators
* Contraindication to magnetic resonance imaging using Gadolinium contrast enhancement (e.g. pacemaker, metallic implant or impaired renal function)
* Rapid extracranial disease progression that in the opinion of the investigators confer a high risk of drop out from the study without evaluation scan at 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-08-20 (Estimated); Study Completion 2023-08-20 (Estimated)

PRIMARY OUTCOMES:
Freedom from progression of treated metastasis | 3 months post treatment
  Freedom from progression of lesion size defined as stable or decreasing unidimensional measurement (longest diameter) on T1-weighted contrast enhanced magnetic resonance imaging (MRI)

SECONDARY OUTCOMES:
Adverse events | 12 months
  Adverse events graded using National Cancer Institute (NCI) Common Toxicity Criteria (CTC) Adverse Events (AE) version 5.0
Overall response | 3 months
  Overall radiographic response of all treated lesions
Neurological status | 6 months
  Neurological status assessed by NANO (neurologic assessment in neuro-oncology) scale
Time to intracranial relapse | From date of treatment until the day of radiologically documented relapse in the brain assessed up to 12 months
  Time to recurrence of treated lesion or occurrence of new lesion(s)
Overall survival | From date of treatment until date of death from any cause assessed up to 12 months
  Overall survival from entry into study
Patient reported outcomes | 6 months
  Health related quality of life measured by the FACT-Br (Functional Assessment of Cancer Therapy - Brain) questionnaire

OTHER OUTCOMES:
Positron emission tomography using fluoro-ethyl tyrosine (FET) tracer before and after treatment | 3 months
  Exploratory endpoint. The measured change in biological tumor volume (BTV) and Tmax/brain (maximal tumor activity) as compared to baseline values.
Dynamic MRI using DCE (dynamic contrast enhancement) perfusion measurement before and after treatment | 3 months
  Exploratory endpoint. The measured change in tumor blood volume measurement, tumor perfusion and tumor permability (Ki) as compared to baseline values.

CONTACTS AND LOCATIONS:
Overall Officials: Søren Møller, MD, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, University of Copenhagen, Copenhagen, Denmark